CLINICAL TRIAL: NCT01008358
Title: Phase II Trial of Anti-CTLA-4 Human Monoclonal Antibody CP-675,206 in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Anti-CTLA-4 Human Monoclonal Antibody CP-675,206 in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-2007-01; EudraCT number 2008-001177-15
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Hepatocellular Carcinoma; Hepatitis C Virus Chronic Infection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: CP 675,206

SUMMARY:
CP-675,206 (tremelimumab) is a fully humanized monoclonal antibody that binds to activated T lymphocytes and by enhancing their activation may produce a stimulation of the immune response against tumoral or viral antigens. In this clinical trial, the ability of tremelimumab to produce tumor responses among hepatitis C virus-infected patients with hepatocellular carcinoma not amenable to other therapies will be explored. Besides, the effect on the replication of the virus will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal diagnosis of HCC
* unresectable disease not amenable to locoregional treatment.
* a 4-week washout period after sorafenib or any other systemic agent
* a 2-month washout period after internal or external radiation
* HCV chronic infection
* Child-Pugh stage A or B
* Measurable disease according to RECIST criteria
* ECOG < 2
* expected survival > 3 months
* Adequate liver, renal and blood functions
* ability to sign informed consent

Exclusion Criteria:

* previous treatment with an anti-CTL-4 agent
* serious infections or disease compromising general health status
* autoimmune disease that requires therapy
* treatment with immunosuppressors
* treatment with investigational agents
* other neoplasms except skin and bladder superficial tumors
* pregnancy or lactation
* SNC metastasis
* HIV infection
* relevant heart disease (NYHA class III or IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Tumor response by Response Evaluation Criteria In Solid Tumors (RECIST)

SECONDARY OUTCOMES:
Changes in Hepatitis C Virus (HCV) viral load

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Prieto-Valtuena, MD, PhD, Study Director — Clinica Universidad de Navarra
Locations (3):
- Spain (3):
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Clinica Universitaria de Navarra, Pamplona

REFERENCES:
- [Derived] Sangro B, Gomez-Martin C, de la Mata M, Inarrairaegui M, Garralda E, Barrera P, Riezu-Boj JI, Larrea E, Alfaro C, Sarobe P, Lasarte JJ, Perez-Gracia JL, Melero I, Prieto J. A clinical trial of CTLA-4 blockade with tremelimumab in patients with hepatocellular carcinoma and chronic hepatitis C. J Hepatol. 2013 Jul;59(1):81-8. doi: 10.1016/j.jhep.2013.02.022. Epub 2013 Mar 4. PMID 23466307